CLINICAL TRIAL: NCT03534583
Title: Alternative Treatments to Help Post Traumatic Stress Disorder
Brief Title: SKY vs. HEP in PTSD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to Covid-19 pandemic related restrictions
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Kamini Vasudev, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111756
Record Dates: First submitted 2018-04-29; First posted 2018-05-23 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Raters, investigators and physicians will not be aware of participant treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Enhancement Program (HEP) (Active Comparator): The Health-Enhancement Program (HEP) is structurally equivalent to a SKY intervention, with similar-sized groups, meeting for 3 consecutive days for 1.5-3 hours. There will then be a a gap of 4 days where participants will practice what they have learned, followed by 3 consecutive days of 1.5-3 hours of instruction. Starting the following week participants will attend once weekly follow up sessions (60-90 min/wk) for 3 weeks and then bimonthly sessions for the next 8 weeks. Participants will be asked to complete 25 min/day of course homework. Participants will learn about health promotion, healthy diet, music, and exercise, but do not learn breathing techniques, or meditation. In HEP, which has been manualized, participants get the support of a group and facilitator, and talk through and try to implement positive health-enhancing life changes, HEP will be delivered by a trained social worker (or equivalent).
  Interventions: Other: Health Enhancement Program
- Sudarshan Kriya Yoga (SKY) (Experimental): The SKY PTSD program is a mind-body resilience building program developed for persons with PTSD. Through SKY breathing, interactive discussions, journaling, yoga and guided meditations, the workshop builds a framework for resilience and empowerment, and develops self-awareness, connectedness and community, and a positive outlook. SKY training will take place in group-format (6-8 participants). During the first week participants will attend three 2.5-3 hour sessions on three consecutive days. There will then be a gap of 4 days where participants can apply the tools provided, followed by three more consecutive days of 1.5-3 hours of instruction. This will be followed by once weekly follow up sessions (90 min/wk) for 3 weeks and then bimonthly sessions (every 2 weeks) for the next 8 weeks. In addition, participants will be asked to practice SKY at home daily (25 min/day) throughout the duration of the study period (up to 26 weeks) and log practice frequency.
  Interventions: Other: Sudarshan Kriya Yoga

INTERVENTIONS:
Other: Sudarshan Kriya Yoga — Participants in the SKY group will undergo an oline 12-week training course conducted by certified teachers of the Art of Living Foundation
  Other Names: SKY
  Arms: Sudarshan Kriya Yoga (SKY)
Other: Health Enhancement Program — Participants in the online HEP will learn about health promotion, healthy diet, music, and exercise, but will not learn breathing techniques, or meditation. HEP will be delivered by trained staff.
  Other Names: HEP
  Arms: Health Enhancement Program (HEP)

SUMMARY:
Post-traumatic stress disorder (PTSD) is the third most common mental illness with a lifetime prevalence rate of 9.2% in Canada. Depression and anxiety are common comorbidities making treatment complex. Currently available treatments for PTSD include medications and talk therapies. However, their best combined response rates are around 50%. Our recent pilot feasibility study showed potential benefits of a breathing based meditation intervention called Sudarshan Kriya Yoga (SKY) in PTSD, as an augmentation treatment. The investigators seek to now assess the safety and efficacy of SKY intervention compared to an active control, Health Enhancement Program (HEP) in a double blind randomized controlled trial. The investigators will include PTSD patients with a wide range of trauma experience including road traffic accidents, childhood, physical, emotional or sexual abuse, or recurrent traumas over the lifespan. Patients will be offered a 12-week program of either SKY or HEP interventions as an add-on to their existing treatment schedules. This study will examine if patients with PTSD experience a reduction in PTSD symptoms from baseline to 12-week follow-up, as measured by the PCL-5 after receiving either HEP or SKY.

DETAILED DESCRIPTION:
STUDY DESIGN: Single-center, blinded (rater, investigator, and clinician), longitudinal, RCT comparing a 12-week SKY online intervention group to a 12-week HEP online intervention group.

STUDY RECRUITMENT: Participants include men and women (n=130), 18-75 years of age, with PTSD. The study will recruit via referrals from the General Adult Ambulatory, the Traumatic Stress Services Program (TSS), the PTSD clinical research unit and the Geriatric Mental Health Program of London Health Sciences Centre at an expected rate of approximately 1 to 2 participants per week. Referred participants will be individuals who in the opinion of investigators or referring physicians will likely meet inclusion and exclusion criteria. A letter will be sent to primary care physicians in London, ON and surrounding area requesting the referral of potential participants. The letter will be accompanied by a poster advertising the study and by a list of the studies inclusion/exclusion criteria. Posters will also be placed online on the websites of the studies investigators as well as websites and social media sites of relevant organizations such as Project Trauma Support and Ivegotyourback911. Online posters will indicate that individuals should not share or comment on posters to protect their identity. Printed posters will be placed in community centres, libraries, hospitals, medical centres, locations where veterans frequent, and locations where first responders work such as fire halls and police stations. Information sessions will be held at locations where first responders work or may frequent to inform potential participants about the study.

SCREENING AND INITIAL ASSESSMENT: Referred potential participants will be provided with a Letter of Information (LOI) to review and consider. Participants will be given a minimum of 24 hours to review the LOI before being contacted over-the-phone by one of the study Research Assistants (RA). During this initial phone call the RA will answer any questions the potential participants have, briefly explain the study, and invite potential participants to a screening appointment to be conducted either remotely or in person. During the initial screening appointment participants will complete the informed consent process which includes an opportunity to ask any questions. Participants will be screened for inclusion and exclusion criteria by a trained member of the research team. These participants will have clinically diagnosed PTSD, further confirmed through a structured clinical interview, the Clinician-administered PTSD Scale for DSM5-past month version (CAPS5). Any additional diagnoses will be screened by the MINI (Mini International Neuropsychiatric Interview). The CAPS5 will also be used to rule out severe depersonalization and derealization as per exclusion criteria. If the participant is above the age of 65 years of age, they will complete a cognitive screening test using the Mini Mental State Examination, MMSE>24 to rule out significant cognitive impairment. Participants meeting all study criteria who wish to join the study will be enrolled and assigned a unique study identifier e.g. HEPSKY001.

RANDOMIZATION: Participants meeting inclusion criteria will be randomized to either SKY or HEP with equal probability (1:1), stratified by gender, using computer generated randomisation numbers. Concealment of randomisation to outcome assessors and investigators will be ensured by an independent consultant who will perform the randomization. The independent consultant will be responsible for randomization and will inform an unblinded study team member of allocation codes. The unblinded study team member will send an email to study participants informing them of their treatment allocation.

TRIAL INTERVENTIONS: The investigators will offer the two interventions, online via Cisco WebEx, in groups of 6-8 participants on a rolling basis 1. Sudarshan Kriya Yoga (SKY): 1. Participants in the SKY group will undergo a 12-week training course conducted by certified teachers of the Art of Living Foundation. 2. HEP Intervention: Participants in HEP will learn about health promotion, healthy diet, music, and exercise, but will not learn breathing techniques, or meditation. HEP will be delivered by trained staff.

All participants will continue to receive standard care through their providers.

STATISTICAL ANALYSIS PLAN: All statistical analyses will be run with the level of statistical significance set at 0.05. Independent samples t tests (for continuous variables) or chi-squared analyses (for categorical variables) will be used to identify whether any differences in demographic or clinical characteristics exist between patients assigned to SKY and HEP. Any variables showing statistically significant differences will be controlled for in the analyses, and sub-group analyses will be completed, as appropriate, to estimate the effect of various demographic or clinical variables. For our Primary Objective 1, the change in PCL-5 scores from baseline to 12-week follow-up of patients assigned to SKY and HEP will be compared using linear mixed models. This approach will account for the clustering of observations since both SKY and HEP will be delivered in a group setting. We will evaluate whether a greater proportion of patients assigned to SKY, compared to HEP, respond to treatment (decrease of at least 10 points on the PCL-5), or go into remission (defined as a PCL-5 score <33), using generalized linear mixed models. In evaluating our Secondary Objectives; depressive symptoms, anxiety, and quality of life, the change score for each measure from baseline to 12-week follow-up of patients assigned to SKY and HEP will be compared using linear mixed models. In evaluating our Exploratory Objectives, linear mixed models will also be used to evaluate the change in levels of inflammatory markers and HF-HRV from baseline to the 12-week follow-up. Correlation analyses will be used to evaluate whether improvement in PCL-5 scores is associated with greater improvement in levels of inflammatory markers and HR-HRV. Lastly, we will evaluate whether the effects found at the 12-week follow-up are maintained at six months. The above analyses (linear mixed models and generalized linear mixed models) will be repeated for PTSD symptoms, depressive symptoms, anxiety and quality of life, comparing scores at baseline and six-months.

Interim analysis may be completed in order to meet one or more of these conditions a) sponsor reporting requirements and/or b) research training requirements of residents and/or c) data safety monitoring board meetings for stop or continue decisions. Prior research ethics board approval will be sought before any interim analysis is conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Between the age of 18 and 75.
2. Has confirmed Axis 1 diagnosis of PTSD as per CAPS5
3. Sufficiently able to hear allowing them to follow verbal instructions. Able to communicate sufficiently in English.
4. Able to sit without physical discomfort for 60 minutes.
5. Willing and able to attend 6 initial SKY training sessions and 75% of follow up sessions.
6. Not pregnant and willing to remain not pregnant for the Duration of the study.
7. Access to a device with a camera and microphone, internet access, and a private space large enough to accommodate a yoga mat (a yoga mat is not required a comfortable floor space or blanket can be substituted).

Exclusion Criteria:

1. Currently participating in other studies on PTSD treatment.
2. Score severe or extreme on Depersonalization (item 29) or Derealization (item 30) of CAPS5.
3. Have other significant mental health diagnosis including bipolar disorder, Schizophrenia, Neurocognitive disorder, and/or severe Personality Disorder (confirmed by Psychiatrist and MINI).
4. Have significant substance dependence, or for those that have significant substance use disorder (have been regularly using within 6 weeks prior to commencement of intervention) or are unable to attend the intervention and assessment sessions while not under the influence of a substance.
5. Have a risk of suicide as elicited by clinical interview (MINI).
6. Have psychotic episodes within the past 12 months.
7. Have a Traumatic Brain Injury (TBI) as defined by loss of consciousness for more than 20 minutes and/or Glasgow Coma Scale score less than or equal to 12.
8. Non-professionals with complex PTSD. Professionals include those who have served in the Canadian armed forces, are public safety personnel or are health care professionals.
9. Currently practice any type of formal meditation, mindfulness or breathing techniques regularly.
10. Have serious cardiovascular disease in the past 12 months (i.e.myocardial infarction, stroke, uncontrolled hypertension or TIA), or a past history of neurological disease (including Parkinson's Disease), seizures, or diabetic neuropathy.
11. Major surgery within 8 weeks prior to commencement of the intervention, or a scheduled major surgery during the intervention period.
12. Have mental health difficulties that has prevented participant from leaving the house, and/or missed appointments in last 3 months.
13. Have vacation plans that will interfere with participant's ability to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-05-29 (Actual)

PRIMARY OUTCOMES:
Change in Post traumatic stress disorder check list (PCL-5) | Change from baseline to weeks 4, 8, 12 and 26.
  The PCL-5 is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. Participants will be asked to rate how bothered they have been by each item in the past month on a 5-point Likert scale ranging from 0-4. Items are summed to provide a total score ranging from 0 to 80, with higher scores indicating more severe symptoms of PTSD.

SECONDARY OUTCOMES:
Change in Hamilton Depression Scale (HAMD-17) | Change from baseline to weeks 4, 8, 12 and 26.
  The HAMD-17 is a 17 item rater administered questionnaire that assesses the severity of the participants depression over the previous two weeks. Scores range from 0 to 50. Higher scores indicated more severe depression.
Change in Beck's Depression Inventory (BDI) | Change from baseline to weeks 4, 8, 12 and 26
  The BDI is a self rated measure of participants depression. The scale consists of 21 questions each with scores ranging from 0 to 3. Total scores range from 0 to 63, with higher scores indicating more severe depression.
Change in Hamilton Anxiety Scale (HAM-A) | Change from baseline to weeks 4, 8, 12 and 26.
  The rater administered HAM-A measures anxiety. The 14 item questionnaire results in a score range of 0 to 56 with higher scores indicating greater anxiety.
Change in Toronto Side Effects Scale (TSES) | Change from baseline to weeks 4, 8, 12 and 26
  The 32 item TSES measures side effects by asking participants to rate both the frequency and severity of each item. An intensity score for each item is calculated by multiplying the frequency by the severity. Higher scores indicate more severe side effects.
Change in World Health Organization Quality of Life Scale (WHOQOL-Bref) | Change from baseline ato weeks 4, 8, 12 and 26
  The WHOQOL-Bref is a self-rated 26-item questionnaire that assess a participants quality of life. Scores are calculated for questions 1 and 2 and the four domains; physical health, psychological, social relationships and environment. A transformed score rates each of the 4 domains from 0 to 100 with higher scores indicating an improved quality of life.
Change in heart rate | Change from baseline to week 12 and week 26.
  Heart rate will be measured using an electrocardiogram (ECG).
Change in Mean Diastolic Blood Pressure as measured by plethysmograph. | Change from baseline to week 12 and week 26.
  Blood pressures will be obtained manually using a standard plethysmograph by a trained research staff. Three manual blood pressures will be recorded at each time point (0, 12, and 26 weeks), from which the change in mean diastolic blood pressure will be computed.
Change in Mean Systolic Blood Pressure as measured by plethysmograph. | Change from baseline to week 12 and week 26.
  Blood pressures will be obtained manually using a standard plethysmograph by a trained research staff. Three manual blood pressures will be recorded at each time point (0, 12, and 26 weeks), from which the change in mean systolic blood pressure will be computed.
Change in blood levels of C- Reactive Protein (CRP). | Change from baseline to week 12 and week 26.
  Enzyme-linked immunosorbent assay (ELISA) will be used to assess blood levels of C- Reactive Protein (CRP).
Change in Heart Rate Variability (HRV). | Change from baseline to week 12 and week 24.
  Heart rate variability (HRV) will be measured using an electrocardiogram (ECG). HRV, will be calculated by standard deviation of all R-R intervals (SDNN) on ECG, root-mean square of successive differences (RMSSD), and number of R-R intervals differing by >50 m sec from adjacent intervals (NN50) in time domain analysis.
Change in blood levels of Interleukin-6 (IL-6) | change from baseline to week 12 and 24.
  ELISA will be used to assess blood levels Interleukin-6 (IL-6)
Change in blood levels of malondialdehyde (MDA) | Change from baseline to week 12 and week 24.
  ELISA will be used to assess blood levels of malondialdehyde (MDA).
Change in blood levels of total antioxidant capacity | Change from baseline to week 12 and week 24.
  ELISA will be used to assess blood levels of total antioxidant capacity (including glutathione)
Change in blood levels of glutathione | Change from baseline to week 12 and week 24.
  ELISA will be used to assess blood levels of glutathione.

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, LHSC, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No